CLINICAL TRIAL: NCT00942656
Title: Effect of Trans Fatty Acids From Ruminant Sources on Risk Factors for Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: David J. Baer, Ph. D., Principal Investigator, USDA-ARS
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 2006-293
Record Dates: First submitted 2009-07-17; First posted 2009-07-21 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Cardiovascular Disease
Keywords: trans fatty acids; ruminant; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Alkalies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: PHVO — base diet plus 3.0% energy mixed isomers of trans fatty acids from partially hydrogenated vegetable oil
Other: CLA — base diet plus 1.0% energy added from cis-9, trans-11 conjugated linoleic acid
Other: VA — base diet plus 3.0% energy added from vaccenic acid
Other: base — base diet containing approximately 0.1% energy of mixed trans fatty acid isomers

SUMMARY:
The objectives of this study are to : 1) determine if vaccenic acid (trans-11-octadecenoic, a naturally occurring trans fatty acid isomer from ruminant animal products) raises LDL cholesterol in a quantitatively comparable manner as mixed trans fatty acid isomers from partially hydrogenated vegetable oils at 3% of energy intake, 2) determine if cis-9, trans-11 conjugated linoleic acid (a naturally occurring polyunsaturated fatty acid from ruminant animal products) raises LDL cholesterol compared to a control diet, and 3) demonstrate that mixed trans fatty acid isomers from partially hydrogenated vegetable oil raises LDL cholesterol compared to a low trans fatty acid diet.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 38 kg/m2
* Age 25 to 65 years during the intervention
* Fasting glucose < 126 mg/dl
* Blood pressure < 160/100 mm Hg (controlled with certain medications)
* Total plasma cholesterol < 280 mg/dl
* Fasting triglycerides < 300 mg/dl

Exclusion Criteria:

* Use of prescription or over-the-counter medications or supplements that alter lipid metabolism.
* History or presence of kidney disease, liver disease, gout, certain cancers, thyroid disease, gastrointestinal, other metabolic diseases, or malabsorption syndromes.
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin.
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets).
* Women who have given birth during the previous 12 months, pregnant women, women who plan to become pregnant or who become pregnant during the study or lactating women.
* Volunteers who routinely participate in heavy exercise or volunteers who initiate an exercise program during the study.
* Volunteers who have lost 10% of body weight within the last 12 months or who plan to initiate a weight loss program during the next 10 months.
* Use of prescription or over-the-counter antiobesity medications or supplements (e.g., phenylpropanolamine, ephedrine, caffeine, during and for at least 6 months prior to the start of the study) or history of a surgical intervention for obesity.
* Active cardiovascular disease (such as heart attack or procedure within the past three months or participation in a cardiac rehabilitation program within last three months, stroke or history/treatment for transient ischemic attacks in the past three months, or documented history of pulmonary embolus in past six months).
* Smokers or other tobacco users (during the 6 months prior to the start of the study).
* Unable or unwilling to give informed consent or communicate with study staff.
* Self-report of alcohol or substance abuse within the past twelve months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion).
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David J Baer, Ph. D., Principal Investigator — United States Department of Agriculture (USDA)
Locations (1):
- USDA-ARS, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

REFERENCES:
- [Derived] Gebauer SK, Destaillats F, Dionisi F, Krauss RM, Baer DJ. Vaccenic acid and trans fatty acid isomers from partially hydrogenated oil both adversely affect LDL cholesterol: a double-blind, randomized controlled trial. Am J Clin Nutr. 2015 Dec;102(6):1339-46. doi: 10.3945/ajcn.115.116129. Epub 2015 Nov 11. PMID 26561632